CLINICAL TRIAL: NCT03047954
Title: Multicentre, Randomised, Double Blind, Placebo-controlled Study of the Efficacy and Safety of Broncho-Vaxom (OM 85 BV) in Children Suffering From Atopic Dermatitis
Brief Title: Broncho-Vaxom (OM 85 BV) in Children Suffering From Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BV-2002/1
Record Dates: First submitted 2017-01-13; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Broncho-Vaxom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Broncho-Vaxom (Experimental): 1 capsule (3.5 mg) per day, administered over 9 months
  Interventions: Drug: Broncho-Vaxom
- Placebo (Placebo Comparator): Matching placebo capsule
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Drug: Broncho-Vaxom — BV is an orally administered immunostimulating preparation, which consists of a lyophilised bacterial extract prepared from 8 bacterial species (Haemophilus influenzae, Streptococcus pneumoniae, Klebsiella pneumoniae and ozaenae, Staphylococcus aureus, Streptococcus pyogenes and viridans, Neisseria catarrhalis)
  Other Names: Imocur; Broncho-Munal; Ommunal; Paxoral; Vaxoral
  Arms: Broncho-Vaxom
Drug: Placebo - Cap — Matching Placebo capsule administered
  Arms: Placebo

SUMMARY:
The objective of this pilot double-blind study was to evaluate the efficacy and the safety of Broncho-Vaxom 1 capsule (3.5 mg) per day for 9 months compared to placebo on the evolution of the disease in children suffering from Atopic Dermatitis (AD).

DETAILED DESCRIPTION:
Children outpatients of both sexes, aged 6 months to 7 years, with AD confirmed by Haniffin-Rajka or Williams et al, and an AD score (SCORAD) between 25 and 70 were included and followed for 9 months. Patients were randomized to receive either Broncho-Vaxom 1 capsule (3.5 mg) per day or the corresponding placebo over 9 months.

Children under general corticotherapy within one month of study start, patients with immunodeficiency, patient's affected body surface area less than 15% or greater than 70% or with known allergy to desonide were excluded.

Outcome measures were a comparisons between the two groups in the number of AD flares during the study after the first month of treatment. Secondary outcome measures were comparisons between the two groups based on SCORAD evolution, area of eczema, amount of corticoids used and parents/investigator assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children aged 6 months to 7 years (in eighth year of life)
* Children with Atopic Dermatitis (Hanifin-Rajka or Williams et al criteria) with affected body surface area ≥15% and ≤ 70%
* 25 ≤ SCORAD ≤ 70
* Written informed consent obtained from the parents/legal Guardian (and the child if applicable)

Exclusion Criteria:

* Children under general corticotherapy within one month of study start
* Children with immunodeficiency
* Children with malignant disease
* Children with SCORAD<25 or >70
* Children with affected body surface area < 15% or >70%
* Children with autoimmune disease
* Children under immunosuppressive or immunostimulating therapy within 1 month of study start
* Children whose parents or Guardians are unable to comply with the requirements of the protocol e.g.completion of patient's diary card
* Children with a known allergy or previous intolerance or known hypersensitivity to the trial drug or any of the corticoids used
* Participation in another clinical trial and/or treatment with an experimental drug within 3 months of study start and during present trial

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 179 (Actual)
Dates: Start 2003-07; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of Atopic Dermatitis (AD) flares over 9 months of treatment | 9 months
  Comparison between experimental and Placebo arms in the number of AD flares

SECONDARY OUTCOMES:
SCORAD Evolution over 9 months of treatment | 9 months
  Comparison between experimental and Placebo arms in SCORAD evolution over 9 months of treatment
Area of eczema involvement | 9 months
  Comparison between experimental and Placebo arms in eczema involvement by measurement and recording of total body surface area affected at 3 monthly intervals as compared with baseline
Amount of corticosteroids used | 9 months
  Comparison between experimental and Placebo arms in amount of corticosteroids used

OTHER OUTCOMES:
Incidence of treatment emergent adverse events | 9 months
  measurement of vital signs, results of physical examinations, number and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yves De Prost, MD, Principal Investigator — Hopital Necker-Enfants Malades

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams HC, Burney PG, Hay RJ, Archer CB, Shipley MJ, Hunter JJ, Bingham EA, Finlay AY, Pembroke AC, Graham-Brown RA, et al. The U.K. Working Party's Diagnostic Criteria for Atopic Dermatitis. I. Derivation of a minimum set of discriminators for atopic dermatitis. Br J Dermatol. 1994 Sep;131(3):383-96. doi: 10.1111/j.1365-2133.1994.tb08530.x. PMID 7918015
- [Background] Wolkerstorfer A, de Waard van der Spek FB, Glazenburg EJ, Mulder PG, Oranje AP. Scoring the severity of atopic dermatitis: three item severity score as a rough system for daily practice and as a pre-screening tool for studies. Acta Derm Venereol. 1999 Sep;79(5):356-9. doi: 10.1080/000155599750010256. PMID 10494710
- [Background] Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology. 1993;186(1):23-31. doi: 10.1159/000247298. PMID 8435513
- [Background] Hanifin JM, Rajka G. Acta Derm Venereol Suppl (Stockh) 1980; 92:44-7